CLINICAL TRIAL: NCT02908204
Title: Long-term Outcomes After Treatment for Superficial Esophageal Squamous Cell Carcinoma
Brief Title: Long-term Outcomes of Superficial Esophageal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Tongji Hospital (Other); The affiliated Hospital of Shihezi University (Unknown)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Other Study IDs: SGZAHGX
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Esophageal Neoplasms
Keywords: superficial esophageal squamous cell carcinoma; efficacy; survival
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endoscopic treatment: Patients underwent endoscopic treatment including Endoscopic Mucosal Resection (EMR), Endoscopic Submucosal Dissection (ESD), Multiband Mucosectomy (MBM), Endoscopic Mucosal Band Ligation(EMBL) and so on.
- Traditional surgery: Patients underwent traditional surgery

SUMMARY:
Tumor is the primary public health problem and the incidence of esophageal cancer showed the increasing trend in the past thirty years. According to the statistics in 2015, the new onset of esophageal cancer is about 477,900 yearly. The mainly pathologic type of esophageal cancer in China is esophageal squamous cell carcinomas, which accounts for more than 90% of patients in China. With the development of endoscopic technics, more and more patients choose to receive the endoscopic procedure rather than traditional surgery. However, the long-term efficacy and outcomes of patients with superficial esophageal squamous cell carcinoma received different interventions remained unclear. Thus, investigators aim to conduct a multi-center retrospective study to investigate the long term outcomes of superficial esophageal squamous cell carcinoma patients receiving endoscopic treatment and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients received endoscopic treatment because of the superficial esophageal disease and had the pathologic diagnosis of squamous cell carcinoma.

Exclusion Criteria:

* Combined with other severe disease
* With a history of esophageal surgery
* Combined with other malignant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with superficial esophageal squamous cell carcinoma underwent endoscopic treatment or traditional surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years after treatment

SECONDARY OUTCOMES:
Recurrence rate | 3 years after treatment
Short-term complications incidence rate | 30 days after treatment
Long-term complications incidence rate | 3 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No